CLINICAL TRIAL: NCT03661463
Title: A Randomised Controlled Trial of Aspirin Versus no Treatment to Reduce Aneurysm Wall Inflammation in Unruptured Intracranial Aneurysms.
Brief Title: Unruptured Intracranial Aneurysm Aspirin Trial (UIAAT).
Acronym: UIAAT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RHM NEU 0341
Record Dates: First submitted 2018-07-12; First posted 2018-09-07 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-08

CONDITIONS: Intracranial Aneurysm; Inflammation
Keywords: Aspirin; Magnetic Resonance Vessel Wall Imaging
MeSH Terms: conditions — Intracranial Aneurysm; Inflammation | interventions — Aspirin

STUDY DESIGN:
Intervention Model Description: 2 Parallel Arms - one with the intervention (Aspirin 300mg OD), and one with no treatment. 29 patients each arm.
Who Masked: Outcomes Assessor
Masking Description: The assessor of radiological outcomes will be blinded to which arm of the trial patients were randomised to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aspirin (Experimental): Aspirin (Acetylsalicylic Acid [ASA]) tablets, 300mg once a day, for 90 days.
  Interventions: Drug: Aspirin
- No Treatment (No Intervention): No medical treatment

INTERVENTIONS:
Drug: Aspirin — Drug
  Other Names: acetylsalicylic acid
  Arms: Aspirin

SUMMARY:
Does Aspirin reduce inflammation in the walls of unruptured brain aneurysms?

Brain aneurysms are balloon-like outpouchings of a blood vessel resulting from a weakness in the vessel wall. They generally cause no symptoms, but can burst and cause a bleed in the brain, resulting in death or disability. Aneurysms occur in 1 in 30 people, but rarely burst, with 1 in 10,000 people having a brain bleed.

Ideally, aneurysms would be treated before they burst to prevent bleeding in the brain. The two ways of treating aneurysms currently are both risky and invasive, and no medications have been shown to reduce the risk of aneurysms bursting.

Aspirin is one of the most common medications, used worldwide to treat pain, fever and inflammation, and for the prevention of strokes and heart attacks. Its anti-inflammatory properties may be beneficial for patients with aneurysms. We know that the walls of burst aneurysms and aneurysms that are about to burst, are more inflamed than those that do not burst. Therefore, a drug that reduces inflammation may reduce the risk of an aneurysm bursting.

We have designed this study to test whether there is a measurable reduction in inflammation in walls of brain aneurysms.

In this study, participants known to have an aneurysm that is not planned for treatment and has not yet burst, take aspirin daily for three months, and have an MRI scan before and after to look for a reduction in inflammation.

If this study is successful it would be the first step towards developing the first medication to help treat patients with aneurysms, representing a huge advance for the 2.1 million people in the UK with this condition.

DETAILED DESCRIPTION:
The Unruptured Intracranial Aneurysm Aspirin Trial (UIAAT) is a single centre, randomised, single blind, open label trial of 300mg aspirin daily versus no treatment for 3 months. 58 patients with an intracranial aneurysm diagnosed on imaging will be recruited - potential participants will be approached by their consultant neurosurgeon or a member of their direct clinical care team.

Patient interviews will take place at Wessex Neurological Centre to coincide wherever possible with standard appointments. Participants will be screened for eligibility and consented during this interview. Following consent, baseline data will be taken to include participants' baseline characteristics, other medications, and comorbidities.

The patients will then undergo a baseline MRI including VWI imaging, and then be randomised to either the 'aspirin 300mg daily' or 'no treatment' arms.

All participants will then be called by a member of the trial team between days 7 and 21 after being commenced in either arm of the trial, to review any issues with taking the medication if they are on that arm, whether they are using their drug diary, and to check for any adverse reactions or events.

Following three months of their allocated treatment, patients will undergo a second, identical MRI scan, to assess whether there is any reduction in the inflammation in the vessel walls of the aneurysms. Patients will be reviewed at this time with their drug dairy, for drug reconciliation and recording of any adverse events. This will be the end of their participation in the trial.

The study topic and design was discussed at a meeting to set research priorities advertised via the Wessex Subarachnoid Haemorrhage group that was convened by a consultant neurosurgeon and a subarachnoid haemorrhage specialist nurse with patients with unruptured and ruptured aneurysms and their carers. At this meeting the investigators clearly identified that it would be beneficial for more research into medical treatments for unruptured aneurysms and felt that with the evidence that the group would be happy to undergo the main two items required for participation in the study - treatment with aspirin and increased scanning frequency and were very supportive of the study design. Indeed the group saw the additional scanning as a strong attraction to participating in the study.

ELIGIBILITY:
Inclusion Criteria:

Participants who will be eligible for inclusion in the study will:

* Have a saccular unruptured intracranial aneurysm identified on imaging (CT, MRI or DSA),
* Aneurysm ≥5mm
* Be aged 18 or over
* Male or female
* Capable of giving written informed consent
* Females of childbearing potential must have a negative pregnancy test. Patients of childbearing potential must agree to use an effective birth control method to avoid pregnancy for the duration of the study.

Exclusion Criteria:

Participants will be ineligible for inclusion in the study if they have any of the following:-

* aneurysms smaller than 5mm in size.
* Aneurysm types of the following nature:

  * Fusiform aneurysms
  * Dissecting aneurysm
  * Traumatic aneurysms
  * Cavernous aneurysms
  * Thrombosed aneurysm
* MRI contraindications:

  * Metallic implant
  * Contrast allergy
  * Claustrophobia
* Aspirin contraindications (or increased risk):

  * Peptic ulceration
  * Bleeding disorder
  * Haemophilia
  * Previous peptic ulceration
  * Severe cardiac failure
  * Severe hepatic dysfunction
  * Severe renal failure
  * Allergy to aspirin or NSAIDs
  * Pregnancy
  * Breastfeeding
  * Alcoholism
  * Steroid usage
  * Severe asthma
  * Gout
* Current warfarin or other anticoagulant use
* Current aspirin or clopidogrel use
* Current NSAID use more than once a month
* Planned treatment of the aneurysm within 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2019-10-24 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
A reduction in aneurysm wall inflammation as measured by MRI vessel wall imaging (VWI). | 3 months
  A reduction in aneurysm wall enhancement index of at least 20% on MRI vessel wall imaging (VWI) at the end of 3 months of aspirin 300mg daily treatment, compared to no treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Diederik Bulters, FRCS (SN), Principal Investigator — Wessex Neurological Centre, Southampton General Hospital, University Hospital Southampton NHS Foundation Trust
Locations (1):
- University Hospital Southampto NHS Foundation Trust, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No